COMIRB APPROVED For Use 05-Sep-2019 20-Aug-2020

Principal Investigator: Anthony Elias, MD

COMIRB No: 16-1001

Version Date: August 27, 2019

Study Title: Phase II trial of fulvestrant plus enzalutamide in ER+/ Her2- advanced

breast cancer

You are being asked to be in a research study. This form provides you with information about the study. A member of the research team will describe this study to you and answer all of your questions. Please read the information below and ask questions about anything you don't understand before deciding whether or not to take part.

# Why is this study being done?

This study plans to learn more about a combination of drugs called fulvestrant and enzalutamide and how they work together to treat your type of cancer. Fulvestrant is a standard treatment for your type of cancer. It works by blocking a hormone receptor on the cancer cells. Enzalutamide has been approved to treat other types of cancer and works to block a different hormone receptor. This study is looking at whether the two drugs can work together to help prevent the growth of cancer cells better than each drug could by itself.

You are being asked to be in this research study because you have ER+/ Her2- breast cancer that has spread to other areas of your body and you are a candidate for treatment with fulvestrant.

Throughout the rest of this consent form when referenced together, fulvestrant and enzalutamide will be called the "study drugs".

# Other people in this study

Up to 45 people from your area and around the country will participate in this study.

# What happens if I join this study?

If you join the study, you will be asked to sign this consent form before you receive any study related tests or procedures. You will be given a copy of this form to keep and the original form will be kept at the clinic. Some of these procedures are the same as you would receive as standard of care treatment even if you did not take part in this trial. You can withdraw from the study at any time and this will not affect the standard medical care you receive.

There are three main parts to this study:

- 1. Screening (before treatment)
- 2. Treatment (during the study)
- 3. Follow-up (after treatment)

Page 1 of 14 Initials\_\_\_\_\_

COMIRB 16-1001 PI: Anthony Elias, MD Version Date: 08/27/2019

There are also <u>optional</u> parts of this study. These optional procedures are voluntary and are not required. You can still take part in the main study if you choose not to take part in the optional study procedures.

This next section is an overview of what will be expected of you, and what you can expect if you take part in this study.

# Study visits and procedures

While you are taking part in this study, many of the tests and procedures that will be performed are standard of care for your disease. Some "research" procedures are performed just for this study and are identified below. This study also has both required and optional procedures, which will be listed here.

# Screening

(Weeks -4 to -1)

- Sign informed consent **research**
- Review medical history
- Collect archived tumor tissue **research**
- Tumor imaging scan, such as a CT or MRI
- Physical exam
- Review adverse events
- Review medications
- Blood draw:
  - Standard of care tests including complete blood count, blood chemistry, and blood clotting
  - Tumor biomarkers test research
  - Circulating tumor cells test– research
- Urine test for pregnancy if applicable

If you are pre- or peri-menopausal, you will receive injections of goserelin throughout the study as a standard part of treatment for your disease.

### **Treatment**

(Each cycle is 4 weeks long)

# Cycle 1/ Week 1/ Day 1

- Physical exam
- Review adverse events
- Review medications
- Fulvestrant injection (into your muscle). You may have already started this treatment.
- Receive 8 weeks of enzalutamide (pills) **research**. You will take 4 capsules by mouth every day during this study.
- Tumor biopsy research
- Blood draw (if not collected at screening):
  - Standard of care tests including complete blood count, blood chemistry, and blood clotting


- Tumor biomarkers test research
- Circulating tumor cells test research

# Cycle 1/ Day 15

 Fulvestrant injection (into your muscle). Unless you have previously started this treatment.

# Cycle 2/ Week 5

- Physical exam
- Review adverse events
- Review medications
- Fulvestrant injection (into your muscle)
- Tumor biopsy **research**
- Blood draw:
  - Standard of care tests including complete blood count, blood chemistry, and blood clotting
  - Tumor biomarkers test research
  - Circulating tumor cells test- research

# Cycle 3/ Week 9

- Tumor imaging scan, such as a CT or MRI
- Physical exam
- Review adverse events
- Review medications
- Fulvestrant injection (into your muscle)
- Receive 8 weeks of enzalutamide (pills) research
- Blood draw:
  - Standard of care tests including complete blood count and blood chemistry
  - Tumor biomarkers test research
  - Circulating tumor cells test– research

# Cycle 4/ Week 13

The procedures at this visit will be repeated in each successive cycle (every four weeks) as long as you are benefiting. You will continue to receive 8-week supplies of enzalutamide at every other visit as long as you are benefiting. You will also receive tumor imaging scans, such as a CT or MRI, every 8 weeks up to week 49 and then every 12 weeks thereafter until progression.

- Physical exam
- Review adverse events
- Review medications
- Fulvestrant injection (into your muscle).
- Blood draw:
  - Standard of care tests including complete blood counts and blood chemistry
  - Tumor biomarkers test research

# End of Treatment/Progression

Physical exam


- Review adverse events
- Review medications
- Tumor biopsy **optional research**
- Blood draw:
  - Standard of care tests including complete blood count, blood chemistry, and blood clotting
  - Tumor biomarkers test research
  - Circulating tumor cells test– research

# Follow-up

You will be followed 30 days after the last dose of enzalutamide or before initiation of a new antitumor treatment, whichever occurs first. Staff will follow-up with you at a scheduled clinic visit or may contact you by telephone.

# **Optional study procedures**

Here are the <u>optional</u> parts of this study. *Remember, no matter what you decide to do about this <u>optional</u> part of the study, you may still take part in the main study. If you decide to withdraw your consent for the optional parts, you can continue to take part in the main study, unless you withdraw your consent for the main study as well.* 

Following each optional procedure is a statement asking if you want to participate in the optional procedure. Please read the statement and think about your choice. After reading the sentence, please check "Yes" or "No" and initial next to your choice. If you have any questions, please talk to your doctor or nurse.

# Optional consent for biopsy We would like your permission to allow us to take a biopsy of your tumor at the end of the study, when and if it is determined that your disease has progressed. I give my permission for an additional biopsy of my tumor to be taken at the end of study. Yes No Initials Optional Consent for Future Contact We would like your permission to allow us to contact you in the future to inform you about findings from this research and updates on this study on a periodic basis, when available.

Initials

No

I give my permission for my study doctor (or someone he or she chooses) to contact me to inform me about findings from this research and updates on this

study on a periodic basis, when available.

Yes


### 3. Optional Consent for Data and Specimen Banking for Future Research

Dr. Elias would like to keep some of the data, blood and tissue that is taken during the study but is not used for other tests. If you agree, the data and samples will be kept and may be used in future research to learn more about breast cancer. Your samples will be stored in the Breast Cancer Tissue Bank at the University of Colorado Denver. The research that is done with your data and samples is not designed to specifically help you. It might help people who have breast cancer and other diseases in the future. Reports about research done with your data and samples will not be given to you or your doctor. These reports will not be put in your health records. The research using your data and samples will not affect your care.

The choice to let Dr. Elias keep the data and samples for future research is up to you. No matter what you decide to do, it will not affect the care that you will receive as part of the study. If you decide now that your data and samples can be kept for research, you can change your mind at any time and contact your study doctor to let him or her know that you do not want Dr. Elias to use your samples any longer, and they will no longer be used for research. Otherwise, they may be kept until they are used up, or until Dr. Elias decides to destroy them.

When your data and samples are given to other researchers in the future, Dr. Elias will not give them your name, address, phone number or any other information that will let the researchers know who you are.

Sometimes data and samples are used for genetic research (about diseases that are passed on in families). Even if your data and samples are used for this kind of research, the results will not be told to you and will not be put in your health records. Your data and samples will only be used for research and will not be sold. The research done with your data and samples may help to develop new products in the future, but there is no plan for you to be paid.

The possible benefits of research from your data and samples include learning more about what causes breast cancer and other diseases, how to prevent them and how to treat them. The greatest risk to you is the release of your private information. Dr. Elias will protect your records so that your name, address and phone number will be kept private. The chance that this information will be given to someone else is very small. There will be no cost to you for any data or sample collection and storage by Dr. Elias.

Please read each sentence below and think about your choice. After reading each sentence, check "yes" or "no" and initial next to your choice. If you have questions, please talk to your doctor or nurse. Remember, no matter what you decide to do about the storage and future use of your data and samples, you may still take part in the study.


| 1. | I give my permission for my data, blood and tissue to be kept by Dr. Elias and stored in a central tissue bank at the University of Colorado Denver for future use by the study investigators. | | |
|---|---|---|---|
| | ☐ Yes | ☐ No | Initials |
| 2. | . I give my permissions for my data, blood and tissue samples to be used for research about other health problems (for example: causes of heart disease, osteoporosis, diabetes). | | |
| | ☐ Yes | ☐ No | Initials |
| 3. | chooses) to contact me | give my permission for my study doctor (or someone he or she hooses) to contact me to inform me about findings from this research nd updates on this study on a periodic basis, when available | |
| | ☐ Yes | ☐ No | Initials |

At the end of this consent form, you will also be asked to allow information collected from your specimens to be used. You need to agree to have information from these optional procedures to be used, or you cannot take part in these optional study procedures.

# How long will I be on the study?

You will continue to receive treatment with the study drugs as long as you are benefiting or until you have an unacceptable drug-related side effect. There is no maximum duration of this treatment.

# What are the possible discomforts or risks?

As with any study drug, side effects may occur while taking these study drugs. While taking part in this study, and being treated with the study drugs, you will be watched carefully for any side effects. Some side effects may go away after you stop taking the study drug. Some side effects can be long lasting and may never go away or may even lead to death.

You should talk to your study doctor about any side effects or discomfort you may have. The study doctor may give you some medicine that will help with some side effects. The study doctor may also interrupt or discontinue the study drug.

You will be notified by your study doctor of any new side effects seen in other patients that occur during the time you are on the study. This may affect you wanting to continue in this research study.


Discomforts you may experience while in this study include:

# Risks of Study Drugs:

# Enzalutamide:

# Likely:

- Diarrhea
- Nausea
- Vomiting
- Fatigue or weakness
- Headache
- Feeling hot or flushed
- Increase in blood pressure

# Less likely:

- Dizziness
- Memory impairment
- Restless leg syndrome
- Anxiety
- Nose bleeds
- Dry skin
- Itchy skin
- Skin rash

### Rare. but serious:

- Low white blood cell count, which may increase your risk of infection
- Seizures
- Epileptic seizures
- Hallucination

# Fulvestrant:

### Likely:

- Fatigue or weakness
- Pain, including generalized, back, stomach, and injection site pain
- Headache
- Decrease in blood pressure
- · Feeling hot or flushed
- Nausea
- Vomiting
- Constipation
- Diarrhea
- Bone pain
- Sore throat
- Cough

# Less likely:

· Pelvic and chest pain


- Flu-like symptoms
- Fever
- Loss of appetite
- Anemia (low red blood cell count), which may cause tiredness or weakness
- Swelling in the hands and feet
- Joint swelling
- Dizziness
- Difficulty sleeping
- Numbness or tingling in the hands and feet
- Depression
- Anxiety
- Skin rash
- Sweating
- Urinary tract infection

### Rare. but serious:

- Blood clots in your arms or legs that may reach the lungs
- Vaginal bleeding
- Low white blood cell count, which may increase your risk of infection
- Blood clot in the lungs (also known as pulmonary embolism)

# Risks of having blood taken:

In this study, we plan to take about 3-4 tablespoons of blood from you at screening/week 1, week 5, week 9, week 13, and when your disease progresses. You may feel some pain when the needle goes into your vein, and you could have a bruise over the next few days.

### Risks of biopsy:

In this study, we will take 2 or 3 biopsies from you. There are some risks to taking a biopsy. There is a small chance that you could get an infection where the needle goes in. You may also experience redness, swelling, minor bleeding or bruising at the site where the cut was made or the needle inserted. You may experience mild to moderate pain at the site of the needle puncture. There is also a small chance that you could have an allergic reaction to the numbing medicine. After your skin heals up, you may have a small scar where we take the samples.

# Archival tumor tissue:

A section will be taken from tumor tissue samples you may have had in the past. Since this has already been removed from you, there are no additional risks to you.

# Risks of loss of confidentiality:

There is a risk that people outside of the research team will see your research information. We will do all that we can to protect your information, but it cannot be guaranteed.

# Other possible risks include:


The particular treatment or procedures involved in this study may involve risks to the embryo or fetus which are currently unclear. Women of child-bearing potential should avoid getting pregnant while on this study.

This study may include risks that are unknown at this time.

# What are the possible benefits of the study?

This study is designed for the researcher to learn more about your cancer and how the study drugs affect this type of cancer. However, there is no guarantee that your health will improve if you join this study. Also, there could be risks to being in this study. If there are risks, these are described in the section describing the discomforts or risks.

### Are there alternative treatments?

There may be other ways of treating your cancer. You have the following choices available to you:

- Getting treatment or care for your cancer without being in a study.
- Taking part in a different study.
- Get treatment only for your pain and symptoms, but no treatment for the cancer itself.
- You could also choose to get no treatment at all.

You should talk to your doctor about your choices. Make sure you understand all of your choices before you decide to take part in this study. You may leave this study and still have these other choices available to you.

# Who is paying for this study?

This research is being paid for by The University of Colorado Cancer Center and the Department of Defense. The study drug Enzalutamide is furnished without charge by the manufacturer, Astellas.

# Will I be paid for being in the study?

You will not be paid to be in the study.

# Will I have to pay for anything?

There are some medical treatments that you would get for your condition whether you were in this study or not, such as a biopsy or blood draw. You or your insurance will have to pay for these. There are other medical treatments that you will get because you are in this research study. We will pay for those. We will pay for biopsies and blood collection when they are not needed for your normal care. Otherwise, these procedures may be combined and charges will be sent to your insurance. You or your insurer would also be responsible for paying for the study drug, Fulvestrant. However, the study drug, Enzalutamide, is provided without charge by its manufacturer.


# Is my participation voluntary?

Taking part in this study is voluntary. You have the right to choose not to take part in this study. If you choose to take part, you have the right to stop at any time. If you refuse or decide to withdraw later, you will not lose any benefits or rights to which you are entitled.

In addition, you have the right to change your mind at any point and write to the study doctor to not use your samples for research any longer.

If you leave this study, you will still receive your normal medical care. The only medical care that you will lose is the medical care you are getting as part of this study. You might be able to get that same kind of medical care outside of the study. Ask your study doctor.

If there are any new findings during the study that may affect whether you want to continue to take part, you will be told about them.

# Can I be removed from this study?

The study doctor may decide to stop your participation without your permission if the study doctor thinks that being in the study may cause you harm, or for any other reason. You can still receive the study drug, if your doctor thinks that it is safe for you.

If you are taken out of the study, you will still receive your normal medical care.

# What happens if I am injured or hurt during the study?

If you have an injury while you are in this study, you should call Dr. Anthony Elias immediately. His phone number is 720-848-1030 or 303-266-2059.

We will arrange to get you medical care if you have an injury that is caused by this research. However, you or your insurance company will have to pay for that care.

# Who do I call if I have questions?

The researcher carrying out this study is Dr. Anthony Elias. You may ask any questions you have now. If you have questions, concerns, or complaints later, you may call Dr. Elias at 720-848-1030 or 303-266-2059. You will be given a copy of this form to keep.

You may have questions about your rights as someone in this study. You can call Dr. Elias with questions. You can also call the responsible Institutional Review Board (COMIRB). You can call them at 303-724-1055.

A description of this clinical trial will be available on http://www.Clinical Trials.gov, as required by U.S. Law. This Web site will not include information that can identify you. You can search this Web site at any time.


# Who will see my research information?

The University of Colorado Denver (UCD) and its affiliated hospital(s) have rules to protect information about you. Federal and state laws including the Health Insurance Portability and Accountability Act (HIPAA) also protect your privacy. This part of the consent form tells you what information about you may be collected in this study and who might see or use it.

The institutions involved in this study include:

- University of Colorado Denver
- University of Colorado Hospital

We cannot do this study without your permission to see, use and give out your information. You do not have to give us this permission. If you do not, then you may not join this study.

We will see, use and disclose your information only as described in this form and in our Notice of Privacy Practices; however, people outside the UCD and its affiliate hospitals may not be covered by this obligation.

We will do everything we can to maintain the confidentiality of your personal information but confidentiality cannot be guaranteed.

The use and disclosure of your information has no time limit. You can cancel your permission to use and disclose your information at any time by writing to the study's Principal Investigator (PI), at the name and address listed below. If you do cancel your permission to use and disclose your information, your part in this study will end and no further information about you will be collected. Your cancellation would not affect information already collected in this study.

Anthony Elias, MD Mailstop 8117 12801 E. 17<sup>th</sup> Ave. Aurora. CO 80045

Both the research records that identify you and the consent form signed by you may be looked at by others who have a legal right to see that information, such as:

- Federal offices such as the Food and Drug Administration (FDA) and the Office of Human Research Protections (OHRP) that protect research subjects like you.
- People at the Colorado Multiple Institutional Review Board (COMIRB)
- The study doctor and the rest of the study team.
- The Independent Research Monitor, Dr. Elaine Lam, who is responsible for overseeing the safety of this research, and to report observations or findings to the IRB or designated institutional officials.
- Medivation and Astellas, the companies providing the drug, will see only coded information.
- Officials at the institution where the research is conducted and officials at other institutions involved in this study who are in charge of making sure that we follow all of the rules for research.

We might talk about this research study at meetings. We might also print the results of this research study in relevant journals. But we will always keep the names of the research subjects, like you, private.


You have the right to request access to your personal health information from the Investigator.

The investigator (or staff acting on behalf of the investigator) will use your information for the research outlined in this consent form. They will also make all or some of the following health information about you collected in this study available to other sites participating in this study.

# Information about you that will be seen, collected, used and disclosed in this study:

- Name and Demographic Information (age, sex, ethnicity, address, phone number, etc.
- Portions of your previous and current Medical Records that are relevant to this study, including but not limited to Diagnosis(es), History and Physical, laboratory or tissue studies, radiology studies, procedure results
- Research Visit and Research Test records
- Tissue samples and the data with the samples.
- Billing or financial information

# **Genetic Information Nondiscrimination Act (GINA)**

A Federal law, called the Genetic Information Nondiscrimination Act (GINA), generally makes it illegal for health insurance companies, group health plans, and most employers to discriminate against you based on your genetic information. This law will generally protect you in the following ways:

- Health insurance companies and group health plans may not request your genetic information that we get from this research.
- Health insurance companies and group health plans may not use your genetic information when making decisions regarding your eligibility or premiums.
- Employers with 15 or more employees may not use your genetic information that we
  get from this research when making a decision to hire, promote, or fire you, or when
  setting the terms of your employment.

All health insurance companies and group health plans must follow this law by May 21, 2010. All employers with 15 or more employees must follow this law as of November 21, 2009.

Be aware that this new Federal law does not protect you against genetic discrimination by companies that sell life insurance, disability insurance, or long-term care insurance.

# What happens to Data, Tissue, Blood and Specimens that are collected in this study?

Scientists at the University of Colorado Denver and the hospitals involved in this study work to find the causes and cures of disease. The data, tissue, blood and specimens collected from you during this study are important to this study and to future research. If you join this study:

- The data, tissue, blood, or other specimens given by you to the investigators for this
  research no longer belong to you.
- Both the investigators and any sponsor of this research may study your data, tissue, blood, or other specimens collected from you.


- If data, tissue, blood, or other specimens are in a form that identifies you, UCD or the
  hospitals involved in this study may use them for future research only with your
  consent or Institutional Review Board (IRB) approval.
- Any product or idea created by the researchers working on this study will not belong to you.
- There is no plan for you to receive any financial benefit from the creation, use or sale of such a product or idea.

# **HIPAA Authorization for Optional Additional Study Procedures**

In this form, you were given the option to agree to additional, optional research procedures. You must also give us your permission, under HIPAA rules, to use and disclose the information collected from these optional procedures, as described above.

Some of these optional procedures may involve genetic testing or the use of your genetic information. Your genetic information will not be released to others.

If you decline to give us permission to use and disclose your information, you cannot take part in these optional procedures, but you can still participate in the main study. Please initial next to your choice:

| <br>I give permission for my information, from the optional procedures I have agreed to above, to be used and disclosed as described in this section. |
|---|
| I do not give permission for my information for any optional procedures to be used and disclosed; I understand that I will not participate in any optional procedures. |

# Agreement to be in this study and use my data

I have read this paper about the study or it was read to me. I understand the possible risks and benefits of this study. I understand and authorize the access, use and disclosure of my information as stated in this form. I know that being in this study is voluntary. If I choose to be in this study, I will get a signed and dated copy of this consent form.

| Signature: | Date: |
|----------------------------|-------|
| Print Name: | |
| Consent form explained by: | Date: |
| Print Name: | |

If applicable, the signature line for witness is required for consent of non-reading subjects and consent using a short form.


| Witness Signature: | Date: |
|----------------------------|-------|
| Witness Print Name: | |
| Witness of Signature | |
| Witness of consent process | |



# **UCCC Informed Consent Process Documentation**

| COMIRB# | Patient Initials | Subject Number |
|---|---|---|
| Type of ICF (i.e. screening, main, optional) | | |
| Version date:(CIRB = protocol version) | IRB Approval dat<br>(CIRB = ICF versio | |
| The clinical investigator or trained delegate has: | | |

**Initials** Date Thoroughly reviewed the study treatments, procedures, risks, schedules and expenses with the patient and/or legal guardian. Provided adequate opportunity to read the IRB approved consent and HIPAA form. Provided adequate opportunity to consider all options. Exchanged information and responded to questions. Verified understanding of this information. Obtained voluntary agreement to participate in the clinical trial. Verified the date of signature on the consent document. Consent was obtained before the subject began participation in the study. Provided the patient and/or legal guardian with a copy of the consent document that was given to subject to obtain consent. Provided the patient and/or legal guardian with the CCTO Internal Patient Card (If Applicable). If N/A, write N/A next to initials. Retained the original signed consent document in the study This consent form has been sent to Health InforMatics to be added to the participant's medical chart.